CLINICAL TRIAL: NCT00321087
Title: Phase II Efficacy and Safety of Taro Pharmaceuticals' Pro-Drug T2000 (1,3-Dimethoxymethyl-5,5-Diphenyl-Barbituric Acid) In Patients With Essential Tremor: A Randomized, Double-Blind, Placebo-Controlled, Sequential Dose Escalation Study
Brief Title: A Study of T2000 in Essential Tremor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Medical Director, Taro Pharmaceuticals USA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T2000-0533
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Essential Tremor
Keywords: Movement Disorder
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): T2000 dose escalation
  Interventions: Drug: T2000
- 2 (Experimental): Placebo followed by T2000 dose escalation
  Interventions: Drug: T2000
- 3 (Experimental): Placebo followed by T2000 dose escalation
  Interventions: Drug: T2000

INTERVENTIONS:
Drug: T2000 — Dose escalation from 600 to 1000 mg
  Arms: 1
Drug: T2000 — Placebo followed by T2000 dose escalation from 600 to 1000 mg
  Arms: 2
Drug: T2000 — Placebo followed by dose escalation from 600 to 1000
  Arms: 3

SUMMARY:
This study will evaluate the safety and efficacy of T2000 when used to treat patients with moderate to severe essential tremor over a 20 week period.

Essential tremor (ET) is a common form of involuntary shaking not related to Parkinson's disease. The medications that are currently used to treat ET work in a small proportion of patients and provide only partial improvement in symptoms. Use of these current medications is also limited by side-effects in many patients.

T2000 is a medication currently under development for the treatment of essential tremor. Although T2000 is a new medication, it belongs to a class of medications that has been used for many years for the treatment of a variety of medical conditions. In previous studies, T2000 appeared to be effective in controlling symptoms of ET and some patients with severe ET had major improvements in tremor. T2000 was well tolerated for periods up to 20 days and the minimal side-effects seen were those that would be expected for medications in this class.

The current study will evaluate the safety and efficacy of T2000 in patients with moderate to severe essential tremor. Patients will receive doses of T2000 beginning at 600 mg a day, followed by 800 mg a day and up to 1000 mg a day. The total duration of treatment will be 20 weeks. Patient's tremor and neurological examination will be monitored throughout the study. The response to T2000 will be determined by comparing the severity of tremor while patients are receiving T2000 compared to the tremor observed without active medication.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed essential tremor by NIH criteria
* Significant functional activity limitation due to ET
* Patients who have failed, are inadequately treated or cannot tolerate alternative treatments for ET as well as treatment naïve patients who have considered but declined alternative treatment

Exclusion Criteria:

* Patients adequately controlled without side effects on a current ET treatment
* Pregnant patients or patients who may become pregnant during the study
* Patients with other medical conditions that may cause tremor, such as Parkinson's disease or active hyperthyroidism
* Patients taking medications that might produce tremor or interfere with the evaluation of tremor such as CNS-stimulants or beta-blockers
* Patients who must take medications that alter liver metabolism as well as patients with liver disease or coagulation disorders
* Patients with seizure disorders
* Patients with a history of allergy or hypersensitivity reaction to barbiturates or other related medications, such as phenobarbital or phenytoin
* Patient with significant general medical or clinical laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on tremor will be measured by a tremor scale as well as by assessment of functional activity with specific tasks. Patients receiving active treatment will be compared to placebo at 2 months of treatment. | Up to 6 months
Response at various dosages will be compared to baseline for all patients. | Up to 6 months

SECONDARY OUTCOMES:
Safety parameters including neurological examination, blood tests and EKG will be monitored throughout the treatment period and during withdrawal of the medication. | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Investigator Site, London, Ontario
  - Investigator Site, Ottawa, Ontario
  - Investigator Site, Toronto, Ontario